CLINICAL TRIAL: NCT02545257
Title: Development of a Coordinated, Community-Based Medication Management Model for Home-Dwelling Aged in Primary Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Helsinki (Other)
Collaborators: City of Lohja, Services for Aged People (Unknown); Lohjan 1. Apteekki (Other); Social Insurance Institution, Finland (Other)
Responsible Party: Principal Investigator, Terhi Toivo, Project coordinator, MSc (Pharm), PhD student, University of Helsinki
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 153/13/03/00/2015
Record Dates: First submitted 2015-09-04; First posted 2015-09-09 (Estimated); Last update posted 2019-03-12 (Actual); Status verified 2019-03

CONDITIONS: Drug Therapy, Combination; Inappropriate Prescribing; Polypharmacy
Keywords: Aged people; Home care; Drug related problems, DRPs; Coordinated medication management model

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active comparator (Active Comparator): In addition to normal, standard care, participants allocated to intervention group will receive a coordinated medication management model containing prescription review, drug-related problems (DRP) risk assessment and required action based on the DRP risk assessment.
  Interventions: Other: Coordinated medication management model
- Control group (standard care) (No Intervention): Normal, standard care (control group)

INTERVENTIONS:
Other: Coordinated medication management model — Stage I: a prescription review conducted by community pharmacists Stage II: practical nurse-administered Drug-related Problem Risk Assessment Tool Stage III: Required health care action based on the result of the DRP -Risk Assessment Tool
  Arms: Active comparator

SUMMARY:
The objective of this randomized controlled trial is to develop a coordinated, multiprofessional medication management model for home-dwelling aged in primary care and to study the effectiveness of this model. The main hypothesis is that the new model helps to identify aged people having potential risks with their medications and thus allows solving these risks.

DETAILED DESCRIPTION:
The demand for long-term home health care services is increasing due the demographic and societal developments. Aged people needing home care are increasingly older, have many chronic diseases and use multiple medicines and thus, are at high risk for drug-related problems (DRPs). In Finland, national and local healthcare and aged care strategies target to allowing aged people (over 65 years) living in their own homes as long as possible. This minimizes the costs of institutionalized care and also targets to add the quality of life of aged people. New approaches and service models are needed to meet these challenges.

The present study focuses on the development of a coordinated medication management model which aims to ensure the safe medication practises for home-dwelling aged in primary care. In the previous parts of this study project were developed a model for comprehensive medication review process (CMR) and a Drug-Related Problem Risk Assessment Tool. The present study uses a multistage intervention in which medications are reviewed (prescription review) in a community pharmacy using the SFINX-database to identify clinically significant drug-drug interactions and the Salko-database which identifies potentially inappropriate medications for aged people. In the next stage practical nurses use the Drug-Related Problem Risk Assessment Tool to identify potential risks. The following stages are based on the results from the risk assessment tool. Potential options are, e.g.,physician consultation, more frequent home care visits, counselling given by the community pharmacy or comprehensive medication review (CMR). The CMR process is only targeted to a limited group of study participants with clinically significant DRP who probably will benefit from more comprehensive CMR.

ELIGIBILITY:
Inclusion Criteria:

* Home-dwelling over 65 year-old persons receiving regular home care from the City of Lohja

Exclusion Criteria:

* Home care is not given regularly

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 191 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
GDS-15 (Geriatric Depression Scale) | Change from baseline at 12 and 24 months
MMSE (Mini-Mental State Examination) | Change from baseline at 12 and 24 months
  Cognitive ability
MNA (Malnutrition Assessment) | Change from baseline at 12 and 24 months
Time to rise from a chair and return to the seated position 5 times (Lower extremity function). | Change from baseline at 12 and 24 months
Orthostatic hypotension (Short test, Freeman et al. 2011) | Change from baseline at 12 and 24 months
AUDIT-C (Alcohol Use Disorder Identification Test, version C) | Change from baseline at 12 and 24 months
UDI-6 (Urinary Distress Inventory) | Change from baseline at 12 and 24 months
Rava (Functioning and disability, Finnish Consulting Group) | Change from baseline at 12 and 24 months
Potentially inappropriate medicines (PIM) (Clinically significant drug-drug interactions, potentially inappropriate medicines for aged), identified from medication list review chart | Change from baseline at 12 and 24 months
  PIMs are identified with prescription review using SFINX database (clinically significant drug-drug interactions) and Salko database (e.g., for identifying potentially inappropriate medicines for the aged, anticholinergic and serotonergic load).

SECONDARY OUTCOMES:
Use of health care services: visits to physician | at 12 and 24 months from baseline
  Number of visits (previous 3 months)
Use of health care services: hospital days | at 12 and 24 months from baseline
  Number of hospital days (previous 3 months)
Use of health care services: home care services | at 12 and 24 months from baseline
  Services delivered to home (previous 3 months)

CONTACTS AND LOCATIONS:
Overall Officials: Marja SA Airaksinen, Professor, Study Chair — University of Helsinki; Juha T Puustinen, Docent, Study Director — University of Helsinki
Locations (2):
- Finland (2):
  - 1st Pharmacy of Lohja, Lohja
  - Services for aged people, Lohja

REFERENCES:
- [Result] Dimitrow MS, Leikola SN, Kivela SL, Passi S, Lukkari P, Airaksinen MS. Feasibility of a practical nurse administered risk assessment tool for drug-related problems in home care. Scand J Public Health. 2015 Nov;43(7):761-9. doi: 10.1177/1403494815591719. Epub 2015 Jul 7. PMID 26152737
- [Result] Dimitrow MS, Mykkanen SI, Leikola SN, Kivela SL, Lyles A, Airaksinen MS. Content validation of a tool for assessing risks for drug-related problems to be used by practical nurses caring for home-dwelling clients aged >/=65 years: a Delphi survey. Eur J Clin Pharmacol. 2014 Aug;70(8):991-1002. doi: 10.1007/s00228-014-1699-5. Epub 2014 Jun 1. PMID 24879605
- [Result] Dimitrow MS, Airaksinen MS, Kivela SL, Lyles A, Leikola SN. Comparison of prescribing criteria to evaluate the appropriateness of drug treatment in individuals aged 65 and older: a systematic review. J Am Geriatr Soc. 2011 Aug;59(8):1521-30. doi: 10.1111/j.1532-5415.2011.03497.x. Epub 2011 Jul 28. PMID 21797829
- [Result] Bulajeva A, Labberton L, Leikola S, Pohjanoksa-Mantyla M, Geurts MM, de Gier JJ, Airaksinen M. Medication review practices in European countries. Res Social Adm Pharm. 2014 Sep-Oct;10(5):731-40. doi: 10.1016/j.sapharm.2014.02.005. Epub 2014 Feb 24. PMID 24661800
- [Result] Leikola S, Tuomainen L, Peura S, Laurikainen A, Lyles A, Savela E, Airaksinen M. Comprehensive medication review: development of a collaborative procedure. Int J Clin Pharm. 2012 Aug;34(4):510-4. doi: 10.1007/s11096-012-9662-y. Epub 2012 Jun 19. PMID 22711383
- [Result] Leikola S, Dimitrow M, Lyles A, Pitkala K, Airaksinen M. Potentially inappropriate medication use among Finnish non-institutionalized people aged >/=65 years: a register-based, cross-sectional, national study. Drugs Aging. 2011 Mar 1;28(3):227-36. doi: 10.2165/11586890-000000000-00000. PMID 21329402
- [Result] Leikola SN, Tuomainen L, Ovaskainen H, Peura S, Sevon-Vilkman N, Tanskanen P, Airaksinen MS. Continuing education course to attain collaborative comprehensive medication review competencies. Am J Pharm Educ. 2009 Oct 1;73(6):108. doi: 10.5688/aj7306108. PMID 19885077
- [Result] Leikola SN, Virolainen J, Tuomainen L, Tuominen RK, Airaksinen MS. Comprehensive medication reviews for elderly patients: findings and recommendations to physicians. J Am Pharm Assoc (2003). 2012 Sep-Oct;52(5):630-3. doi: 10.1331/JAPhA.2012.10163. PMID 23023843
- [Result] Dimitrow M, Leikola S, Kivela SL, Airaksinen M, Mykkanen S, Puustinen J. [Inappropriate medication use among the aged. Review of the criteria]. Duodecim. 2013;129(11):1159-66. Finnish. PMID 23819202
- [Result] Puustinen J, Lahteenmaki R, Polo-Kantola P, Salo P, Vahlberg T, Lyles A, Neuvonen PJ, Partinen M, Raiha I, Kivela SL. Effect of withdrawal from long-term use of temazepam, zopiclone or zolpidem as hypnotic agents on cognition in older adults. Eur J Clin Pharmacol. 2014 Mar;70(3):319-29. doi: 10.1007/s00228-013-1613-6. Epub 2013 Dec 12. PMID 24337417
- [Result] Puustinen J, Nurminen J, Vahlberg T, Lyles A, Isoaho R, Raiha I, Kivela SL. CNS medications as predictors of precipitous cognitive decline in the cognitively disabled aged: a longitudinal population-based study. Dement Geriatr Cogn Dis Extra. 2012 Jan;2(1):57-68. doi: 10.1159/000336710. Epub 2012 Mar 16. PMID 22619661
- [Result] Puustinen J, Nurminen J, Lopponen M, Vahlberg T, Isoaho R, Raiha I, Kivela SL. Use of CNS medications and cognitive decline in the aged: a longitudinal population-based study. BMC Geriatr. 2011 Nov 1;11:70. doi: 10.1186/1471-2318-11-70. PMID 22044595
- [Result] Nurminen J, Puustinen J, Piirtola M, Vahlberg T, Lyles A, Kivela SL. Opioids, antiepileptic and anticholinergic drugs and the risk of fractures in patients 65 years of age and older: a prospective population-based study. Age Ageing. 2013 May;42(3):318-24. doi: 10.1093/ageing/afs178. Epub 2012 Nov 29. PMID 23204431
- [Result] Puustinen J, Nurminen J, Kukola M, Vahlberg T, Laine K, Kivela SL. Associations between use of benzodiazepines or related drugs and health, physical abilities and cognitive function: a non-randomised clinical study in the elderly. Drugs Aging. 2007;24(12):1045-59. doi: 10.2165/00002512-200724120-00007. PMID 18020536
- [Result] Toivo T, Dimitrow M, Puustinen J, Savela E, Pelkonen K, Kiuru V, Suominen T, Kinnunen S, Uunimaki M, Kivela SL, Leikola S, Airaksinen M. Coordinating resources for prospective medication risk management of older home care clients in primary care: procedure development and RCT study design for demonstrating its effectiveness. BMC Geriatr. 2018 Mar 16;18(1):74. doi: 10.1186/s12877-018-0737-z. PMID 29548304
- [Derived] Toivo T, Airaksinen M, Dimitrow M, Savela E, Pelkonen K, Kiuru V, Suominen T, Uunimaki M, Kivela SL, Leikola S, Puustinen J. Enhanced coordination of care to reduce medication risks in older home care clients in primary care: a randomized controlled trial. BMC Geriatr. 2019 Nov 27;19(1):332. doi: 10.1186/s12877-019-1353-2. PMID 31775650
- See also: Leikola S. Development and Application of Comprehensive Medication Review Procedure to Community-Dwelling Elderly. Doctoral Thesis, University of Helsinki, 2012 — http://urn.fi/URN:ISBN:978-952-10-7698-5
- See also: Puustinen J. Benzodiazepines and Cognitive Functioning in Older Adults. With Emphasis on Long-Term Use and Withdrawal. Doctoral Thesis, University of Turku, 2014 — http://urn.fi/URN:ISBN:978-951-29-5710-1